CLINICAL TRIAL: NCT00752882
Title: Comparison of Ceftazidime Pharmacokinetic in Cerebrospinal Fluid Between Continuous and Intermittent Administration
Brief Title: Ceftazidime Pharmacokinetic in Cerebrospinal Fluid Between Continuous and Intermittent Administration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0025
Record Dates: First submitted 2007-09-13; First posted 2008-09-16 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pseudomonas Aeruginosa Meningitis
Keywords: Ceftazidime; Pharmacokinetics; Pseudomonas; aeruginosa; Meningitis; Patients; hospitalised; cerebrolesion; acquired; pneumopathy; mechanic; ventilation
MeSH Terms: conditions — Pseudomonas Infections; Meningitis; Lung Diseases; Respiratory Aspiration | interventions — Ceftazidime

INTERVENTIONS:
Drug: ceftazidime

SUMMARY:
Meningitis is an infection where morbidity and mortality depend on the delay of the initial treatment for a good prognostic. The antibiotherapy rapidity allows to decrease the mortality. Intermittent administration of ceftazidime is a reference treatment of Pseudomonas aeruginosa meningitis. In the case of Pseudomonas aeruginosa pneumopathy, ceftazidime can be administered by intermittent injections or by continuous perfusion. The continuous administration of ceftazidime is not validated in Pseudomonas aeruginosa meningitis. However, ceftazidime is a time dependant antibiotic and continuous treatment would provide a more efficient therapeutic. The aim of this study is to determine if the continuous administration of ceftazidime could permit a better therapeutic practice of Pseudomonas aeruginosa meningitis compared with intermittent administrations.

DETAILED DESCRIPTION:
This study will compare the administration of ceftazidime by intermittent intravenous injections (29 mg/kg 30min ×3/day) and by continuous infusion (86 mg/kg/24 h, preceded by 29 mg/kg/30 min). The main evaluation criterion of the study is the measure of the time during which ceftazidime concentration is above minimal inhibitive concentration of Pseudomonas aeruginosa in cerebrospinal fluid. This study will be developed in a neurological intensive care department. Inclusion criteria will be essentially, patients aged over 18 years old, hospitalised for a cerebrolesion associated to a hydrocephalus drained by an external ventricular derivation, an acquired pneumopathy under mechanic ventilation since more 7 days in the department of neurological intensive care. This study is a prospective randomised, simple blind and divided in two parts. The first part of the study is a study with parallel group comparing the treatment initiation between a continuous and an intermittent treatment of ceftazidime. The second part of the study is a cross-over study. One patient group will receive a continuous treatment of ceftazidime and the other patient group will receive an intermittent treatment of ceftazidime.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 years old,
* patients hospitalised for a cerebrolesion associated to a hydrocephalus drained by an external ventricular derivation, an acquired pneumopathy under mechanic ventilation since more 7 days in the department of neurological intensive care

Exclusion Criteria:

* patients treated by ceftazidime 15 days before the beginning of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Tarbouriech, Dr, Principal Investigator — University Hospital, Clermont-Ferrand